CLINICAL TRIAL: NCT06441903
Title: Connective Tissue of Pectoralis Major Muscle: Anatomical Study
Acronym: USPEC
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/02
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tendon Injury - Upper Limb
Keywords: Anterior Deltoid Tendon; Anterior Lamina Pectoralis Major; Posterior Lamina Pectoralis Major; Pectoralis Major Tendon; Ultrasound; Deep Fascia Pectoralis Major; Delto Pectoral Tendon
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with no history of pectoralis major
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Through systematic ultrasound visualization of the pectoralis major muscle, we seek to directly visualize and characterize the different intra- and extra-muscular connective structures of the muscle - Delto Pectoral Tendon (DPT) , Distal Pectoralis Major Tendon (PMT), Anterior Deltoid Tendon (ADT), Anterior Pretendinous Lamina of the Pectoralis Major (ALPM), Posterior Pretendinous Lamina of the Pectoralis Major (PLPM) and Deep Fascia of the Pectoral Major (DFPM) - constituting its connective skeleton, with particular attention to its distal portion near the humerus and on the search for this DPT tendon.
  Other Names: Shoulder ultrasound with focus on pectoralis major muscle connective skeleton and distal tendon

SUMMARY:
The delto-pectoral tendon (DPT) is a new tendon recently identified. It completes the insertion of the pectoralis major and perfectly explains the different injuries encountered.

The objective of this observational study is to visualize this new tendon, the DPT, using ultrasound, to measure it, to characterize its role in the overall architecture of the pectoralis major muscle and to analyze its relationship with its main tendon and the anterior and posterior laminae.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years,
* Consultation for a musculoskeletal pathology of the upper limb

Exclusion Criteria:

* History of pathology of the pectoralis major or of the distal tendon of the pectoralis major
* Pregnant or breastfeeding women
* Patient under protection of the adults (guardianship, curators or safeguard of justice)
* Unable to understand
* Opposition by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with no history of pectoralis major and consulting for a musculoskeletal pathology of the upper limb
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Ultrasound visualization of Delto Pectoral Tendon | Day 1

SECONDARY OUTCOMES:
Measurement of DPT by ultrasonography (height, length and thickness in mm) | Day 1
Measurement of ADT by ultrasonography (height, length and thickness in mm) | Day 1
Measurement of PMT by ultrasonography (height, length and thickness in mm) | Day 1
Measurement of the distances in mm between the PMT humeral insertion and the different connective structures: ADT, DPT, ALPM, PLPM and DFPM | Day 1
Ultrasound visualization of the clavicular and sternal portions of the pectoralis major. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Ambroise Paré - Hartmann Private Hospital Group, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No